CLINICAL TRIAL: NCT01482104
Title: A Randomized Controlled Blinded Multi-centre Study of Photodynamic Therapy With Methyl-aminolevulinate Comparing a Simplified Regime With the Approved Regime in Patients With Clinical Low-risk Superficial and Nodular Basal Cell Carcinoma.
Brief Title: New Versus Approved Methyl-aminolevulinate Photodynamic Therapy (MAL-PDT) Regime in Basal Cell Carcinoma (BCC)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Akershus Dermatological Centre (Unknown); Helse Stavanger HF (Other Government); Oslo University Hospital (Other); Førde Central Hospital (Other); Haukeland University Hospital (Other); Hudlegekontoret Lillehammer (Unknown); Hudlegene på Holtet DA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC-004; 2011-004797-28 (EudraCT Number)
Record Dates: First submitted 2011-11-17; First posted 2011-11-30 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-10

CONDITIONS: Skin Neoplasms; Carcinoma, Basal Cell
Keywords: Photochemotherapy; methyl 5-aminolevulinate
MeSH Terms: conditions — Skin Neoplasms; Carcinoma, Basal Cell | interventions — methyl 5-aminolevulinate

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAL-PDT re-treatment (Experimental): 1 treatment of MAL-PDT with re-treatment of non-complete responders
  Interventions: Drug: MAL-PDT re-treatment
- usual MAL-PDT (Active Comparator): 2 MAL-PDT treatments 1 week apart
  Interventions: Drug: usual MAL-PDT

INTERVENTIONS:
Drug: MAL-PDT re-treatment — a schedule of 1 single treatment of Metvix(R)-Photodynamic therapy with re-treatment of non-complete responders by 3 months
  Other Names: Methyl-aminolevulinate
  Arms: MAL-PDT re-treatment
Drug: usual MAL-PDT — schedule of 2 standard Metvix(R)- Photodynamic therapy treatment sessions 1 week apart.
  Other Names: Methyl-aminolevulinate
  Arms: usual MAL-PDT

SUMMARY:
Basal cell carcinoma (BCC) is the most common malignant skin lesion in white adults. It is a slow-growing tumour which despite low metastatic potential may cause significant local tissue destruction and patient morbidity. Methyl aminolevulinate cream plus photodynamic therapy (MAL-PDT) for BCC is currently approved for a procedure using 2 treatment sessions 1 week apart. This procedure is considered quite time- and resource-consuming. Introducing a single treatment session, with a new PDT session for treatment failures after 3 months, might represent an attractive simplification.

This randomised controlled single-blinded multi-centre study primarily aims to compare BCC lesion response rate of two treatment schedules: (a) 1 single treatment of Metvix-PDT with re-treatment of non-complete responders by 3 months, and (b) the usual schedule of 2 standard Metvix(R) PDT treatments 1 week apart.

Secondary objectives are to investigate the treatment response in relation to clinical and histological tumour characteristics such as tumour thickness, subtype and immunohistochemical markers.

ELIGIBILITY:
Inclusion Criteria:

* male/female above 18 years of age
* written informed consent
* 1 or more primary histologically verified BCC, clinically assessed as of either superficial of nodular type

Exclusion Criteria:

* pregnancy
* breastfeeding
* Gorlin's syndrome
* porphyria
* xeroderma pigmentosum
* history of arsenic exposure
* known allergy to MAL
* concomitant treatment with immunosuppressive medication
* physical or mental conditions that most likely will prevent patients attending follow-up sessions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
lesions response rate | 3 years
  Number of lesions in clinical complete response at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Magne Børset, PhD prof, Study Director — Norwegian University of Science and Technology
Locations (9):
- Norway (9):
  - Dept Dermatology, Haukeland University Hospital, Bergen
  - Central Hospital Førde, Førde
  - Hudlegekontoret Lillehammer AS, Lillehammer
  - Akerskus Dermatological Centre, Lørenskog
  - Dept Dermatology, Oslo University Hospital, Oslo
  - Dept Surgery, Oslo University Hospital, Oslo
  - Hudlegen på Holtet, Oslo
  - Dept Dermato-Venereology, Stavanger University Hospital, Stavanger
  - Department of Cancer Research and Molecular Medicine, NTNU, Trondheim